CLINICAL TRIAL: NCT06711341
Title: Investigating The Most Effective Exercise Modality in Knee Osteoarthritis; A RCT
Brief Title: Comparing Exercise Programs for Managing Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Mustafa Alabdallah Alalewy, Principal Investigator, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-15/19
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Knee OA; Osteoarthritis; Osteoarthritis (OA) of the Knee
Keywords: Exercise; Knee Osteoarthritis; Pain; Strength; Whole-Body Vibration
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study is a single-blinded randomized controlled trial. Participants are not blinded to their group assignment. However, the researcher responsible for conducting tests and data collection is blinded to the group assignments to avoid any assessment bias. The researcher who handles randomization and group allocation is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Whole-body Vibration (WBV) Training Group (Active Comparator): Participants undergo WBV training as outlined in the WBV intervention, 3 days per week for 3 weeks. The sessions begin with a duration of 10 minutes in the first week, with the duration increasing each week thereafter. They also perform the home exercises assigned to the Control group on the same days as their PRE sessions.
  Interventions: Device: Whole-body Vibration (WBV) Training
- Progressive Resistance Exercise (PRE) Group (Active Comparator): Participants undergo PRE training as outlined in the PRE intervention, 3 days per week for 3 weeks. The training focuses on strengthening the quadriceps muscles using ankle weights. The load is determined using the DeLorme principle at the start of each week. They also perform the home exercises assigned to the Control group on the same days as their PRE sessions.
  Interventions: Behavioral: Progressive Resistance Exercise (PRE)
- Control Group (Home-Based Exercise) (Active Comparator): Participants perform home exercises three days per week for 3 weeks. The exercises consist of range of motion (ROM) and isometric strengthening exercises as detailed in the intervention section.
  Interventions: Behavioral: Home-Based Exercise

INTERVENTIONS:
Device: Whole-body Vibration (WBV) Training — Participants use the "Compex Winplate," designed specifically for vibration training. The device is set with a frequency of 30 Hz and an amplitude of 4 mm. Participants perform a total of 5 exercises consisting of static and dynamic squat exercises, with a 30-second rest period between sets and between different exercises. The exercises and progression over the weeks are as follows:
  Week 1:
  * Static squat with knees flexed at 30° - 2 sets of 30 seconds each
  * Dynamic squat with knees flexed between 0-60° - 2 sets of 30 seconds each
  * Fingertip-to-sole partial dynamic squat with knees flexed at 30° - 2 sets of 30 seconds each
  * Consecutive weight transfer with knees flexed at 45° - 2 sets of 30 seconds each
  * Single leg static squat with knees flexed at 30° - 30 seconds per leg
  Subsequent Weeks: The duration of each set increases by 10 seconds each week. Each training session includes a 5-minute warm-up and a 5-minute cooldown, consisting of joint motion and muscle stretching exercises.
  Other Names: WBV
  Arms: Whole-body Vibration (WBV) Training Group
Behavioral: Progressive Resistance Exercise (PRE) — Training Duration: Participants undergo approximately 15-20 minute training sessions, 3 days per week for 3 weeks.
  Exercise Regimen: The training focuses on strengthening the quadriceps muscles using ankle weights. The load is determined using the DeLorme principle:
  * At the beginning of each week, the 10-repetition maximum (10RM) is measured.
  * During that week, participants perform their training sets as follows:
    * First set: 50% of 10RM
    * Second set: 75% of 10RM
    * Final set: 100% of 10RM Each training session includes a 5-minute warm-up and a 5-minute cooldown, consisting of joint motion and muscle stretching exercises.
  Other Names: PRE
  Arms: Progressive Resistance Exercise (PRE) Group
Behavioral: Home-Based Exercise — Protocol: Participants receive a printed document with instructions for home exercises and are instructed on how to perform the exercises.
  Training Duration: Sessions are conducted three days per week for 3 weeks.
  Exercise Regimen: The exercises include:
  * Bilateral Quadriceps Isometric Exercise: Participants lie on their backs with a roll below each knee, pressing for 10-second holds, totaling 20 repetitions.
  * Knee Extensions: Participants performed knee extensions while seated, holding each extension for 5 seconds, completing 10 repetitions per leg.
  * Knee Range of Motion (ROM) Exercises: Participants lie face down and alternately bend their knees, completing 10 repetitions.
  Each training session includes a 5-minute warm-up and a 5-minute cooldown, consisting of joint motion and muscle stretching exercises
  Arms: Control Group (Home-Based Exercise)

SUMMARY:
The goal of this clinical trial is to assess and compare the effectiveness of three different exercise modalities-whole-body vibration exercise, progressive resistance exercise, and home-based exercise -in improving quadriceps isometric muscle strength, physical function, balance, knee pain, osteoarthritis symptoms, and overall quality of life in individuals with knee osteoarthritis.

The main questions it aims to answer are:

* How do WBV, PRE, and home-based exercise compare in improving quadriceps strength in people with knee osteoarthritis?
* Which exercise modality leads to the greatest improvements in physical function, balance, knee pain, and quality of life?

Researchers will compare the three exercise regimens to determine which is most effective for improving knee function and relieving osteoarthritis symptoms.

Participants will:

* Engage in whole-body vibration exercise, progressive resistance exercise, or home-based exercise for 3 weeks.
* Undergo assessments before and at the end of the exercise program, including tests for physical function and balance (Timed Up and Go Test, 5x Sit to Stand Test) and questionnaires to evaluate knee osteoarthritis symptoms (WOMAC), quality of life (SF-36), and self-reported knee pain (Numeric Rating Scale).

ELIGIBILITY:
Inclusion Criteria:

1. participants between the ages of 45-70,
2. diagnosed with knee osteoarthritis according to ACR criteria (unilateral or bilateral),
3. having grade 2 or 3 tibiofemoral knee osteoarthritis according to Kellgren-Lawrence staging,
4. having knee pain due to OA for a minimum of 3 months prior to enrollment,
5. patients whose medical treatment is not expected to change during the study period.

Exclusion Criteria:

1. having or had undergone knee surgery,
2. patients unable to walk without support,
3. having musculoskeletal limitations that prevent participation in resistance exercises (contracture, fracture, etc.),
4. other neurological, cardiac, respiratory and systemic diseases that will affect physical activity,
5. currently implementing a regular exercise or physical therapy program specific to knee OA

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps Isometric Muscle Strength | at baseline and 3-weeks
  Quadriceps isometric muscle strength is measured using an Isokinetic dynamometer (CSMI Humac Norm, Stoughton, MA). Measurements are taken in a sitting position with the knee positioned at two angles: 30° and 60° of flexion. For each angle, one trial is performed followed by three real measurements, with the highest peak torque recorded in Newton-meters (Nm). Participants are secured to the dynamometer, and all settings and positions are standardized. Prior to measurements, the device is calibrated, and participants perform a 5-minute warm-up and familiarize themselves with the test procedure. Verbal encouragement is provided during the tests.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) Test (Physical Function and Balance) | at baseline and 3-weeks
  The TUG test assesses lower-extremity function performance, dynamic balance, and fall risk. Participants stand up from a standard chair (43 cm height), walk 3 meters, turn around, walk back to the chair, and sit down. Timing is performed using a chronograph, and one practice trial is conducted before the actual test. The entire walking test is timed in seconds.
Five Times Sit to Stand Test (5xSST) (Physical Function and Balance) | at baseline and 3-weeks
  Five Times Sit to Stand Test (5xSST): The 5xSST evaluates functional lower limb strength, transitional movements, balance, and fall risk. Participants sit on a chair with their back supported, fold their arms across their chest, and then sit and stand five times as quickly as possible without resting their back or legs on the chair. Timing is performed using a chronograph.
Numeric Rating Scale (NRS) (Self-reported Knee Pain) | at baseline and 3-weeks
  Self-reported knee pain is assessed using a 10-cm numeric scale, where 0 indicates no pain and 10 represents maximal pain. Participants rate their most severe pain level experienced over the past week, both at rest and during activity.
WOMAC (Knee Osteoarthritis Symptoms and Function) | at baseline and 3-weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) evaluates symptoms and functional status through 24 questions, rated from 0 (best) to 4 (worst). The index includes five questions on knee pain severity, two questions on stiffness, and 17 questions on physical function limitations.
SF-36 (Quality of Life) | at baseline and 3-weeks
  The Medical Outcomes Short Form 36 (SF-36) assesses health-related quality of life through 36 items rated on Likert scales. Various sub-scores reflect different aspects of health-related quality of life, with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Uludağ University Hospital Physical Medicine and Rehabilitation Clinic, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available due to privacy concerns and the fact that the data collected are not intended for sharing outside of the scope of the study's analysis. Additionally, there are no plans for secondary research involving the data.